CLINICAL TRIAL: NCT04696848
Title: A Phase I Study to Determine the Efficacy and Safety of CKD-516 Tablet Combined With Durvalumab(MEDI4736) in Patient Refractory Solid Tumors
Brief Title: The Efficacy and Safety of CKD516 Combined With Durvalumab in Patient Refractory Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Recruitment difficulty
Sponsor: Tae Won Kim (Other)
Responsible Party: Sponsor-Investigator, Tae Won Kim, Professor, Asan Medical Center
Organization: Asan Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-1485
Record Dates: First submitted 2020-12-23; First posted 2021-01-06 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Colorectal Cancer; Solid Tumor
MeSH Terms: conditions — Colorectal Neoplasms | interventions — N-(4-(3-(1H-1,2,4-triazol-1-yl)-4-(3,4,5-trimethoxybenzoyl)phenyl)thiazol-2-yl)-2-amino-3-methylbutanamide; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CKD-516 plus Durvalumab (Experimental): Stage 1 : dose escalation durvalumab (1500 mg Q4W) plus CKD-516 at dose levels (9, 11, or 13 mg/m2) Stage 2 : durvalumab (1500 mg Q4W) plus CKD-516 at recommended phase 2 dose
  Interventions: Drug: CKD-516 plus Durvalumab

INTERVENTIONS:
Drug: CKD-516 plus Durvalumab — Stage 1 : dose escalation durvalumab (1500 mg Q4W) in combination with CKD-516 at 1 of 3 planned dose levels (9, 11, or 13 mg/m2 twice a week for 3 weeks in each cycle, Q4W).
  Stage 2 : durvalumab (1500 mg Q4W) in combination with CKD-516 at recommended phase 2 dose (twice a week for 3 weeks in each cycle, Q4W).
  Other Names: CKD-516 plus MEDI4736

SUMMARY:
This is a single center, open-label, nonrandomized, Phase 1b, dose-escalation study designed to determine maximum tolerated dose (MTD) of CKD-516 in combination with durvalumab and evaluate the safety and tolerability profile, efficacy of CKD-516 and durvalumab treatment.

DETAILED DESCRIPTION:
Dose Escalation cohort (Stage 1) With traditional 3+3 dose-escalation design, the safety, tolerability, and pharmacokinetics of CKD-516 in combination with durvalumab will be evaluated. Three dose levels of CKD-516 (9, 11, 13 mg/m2) will be investigated in combination with durvalumab 1,500 mg. At each dose level, 3 to 6 patients will be enrolled. After completion of 1 cycle of treatment of all patients in each dose level, decision for enrollment of subjects for next dose level will be decided after review of safety profile by safety review (SRM).

Extension cohort (Stage 2) Stage 2 is an exploratory study for the evaluation of the efficacy of recommended phase 2 dose (RP2D) of CKD-516 in the combination with Durvalumab in patients with specific types of solid tumors (listed below).

Arm 1: Colorectal cancer (CRC) Arm 2: Other cancer (Pancreatic cancer, Cholangiocarcinoma, Stomach cancer, Esophageal cancer)

ELIGIBILITY:
Inclusion Criteria:

Stage 1; Dose escalation cohort:

1. Patients with histopathologically confirmed various tumors including CRC, pancreatic cancer, cholangiocarcinoma, stomach cancer, and esophageal cancer, with measurable or non-measurable disease as determined by RECIST version 1.1, who have progressed despite standard therapy or are intolerant of standard therapy, or for whom no standard therapy exists.
2. Age > 20 years at time of study entry
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
4. Must have a life expectancy of at least 12 weeks
5. Body weight >30 kg
6. Adequate normal organ and marrow function as defined below:

   * Haemoglobin ≥9.0 g/dL
   * Absolute neutrophil count (ANC) 1.5 x (> 1500 per mm3)
   * Platelet count ≥75 x 109/L (>75,000 per mm3)
   * Serum bilirubin ≤1.5 x institutional upper limit of normal (ULN). (This will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician)
   * AST (SGOT)/ALT (SGPT) ≤2.5 x institutional upper limit of normal unless liver metastases are present, in which case it must be ≤5x ULN
7. All patients must provide and FFPE tumor sample for tissue-based IHC staining to determine TIL and other correlatives. Tumor tissue can be either from the primary tumor or metastatic biopsy. If tumor tissue is unavailable, samples should be collected with biopsy before treatment. Archived tumor specimens of ≤3 years are acceptable for IHC.
8. Patients must have a site of disease amenable to biopsy, and be a candidate for tumor biopsy to the institutions' guidelines. Patients must be willing to undergo a new tumor biopsy at screening and during therapy on this study.
9. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. Written informed consent and any locally required authorization obtained from the patient/legal representative prior to performing any protocol-related procedures, including screening evaluations.
10. Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

    * Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
    * Women ≥50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).
11. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

Extension Cohorts (Stage 2)

1. Patients with GI cancers confirmed by histopathology or cytologic examination including CRC, pancreatic cancer, cholangiocarcinoma, stomach cancer, and esophageal cancer.

2~11. same above

Exclusion Criteria:

1. Patients with a history of hypersensitivity to the components of study drugs
2. Prior exposure to any immunotherapy
3. Receipt of the last dose of anticancer therapy (chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies) ≤ 14 days prior to the first dose of study drug (in case of nitrosoureas and/or mitomycin, within 6 weeks before study participation)
4. Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria

   * Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician.
   * Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab may be included only after consultation with the Study Physician.
5. Any concurrent chemotherapy, IP, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable.
6. Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of IP. (in case of VATS and/or ONC surgery, within 2 weeks before study participation)
7. History of allogenic organ transplantation.
8. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

   * Patients with vitiligo or alopecia
   * Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
   * Any chronic skin condition that does not require systemic therapy
   * Patients without active disease in the last 5 years may be included but only after consultation with the study physician
   * Patients with celiac disease controlled by diet alone
9. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring adverse events or compromise the ability of the patient to give written informed consent
10. History of another primary malignancy except for

    * Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of IP and of low potential risk for recurrence
    * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
    * Adequately treated carcinoma in situ without evidence of disease
11. History of active primary immunodeficiency
12. Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B, and hepatitis C.

    * Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients with chronic hepatitis B, confirmed by the presence of anti-HBc, receiving antiviral therapy may be enrolled if the disese is controlled for at least 1 month prior to screening. Controlled hepatitis is defined as serum HBV DNA < 2,000 IU/mL by polymerase chain reaction (PCR). Patients with controlled hepatitis B must remain on antiviral therapy, per institutional practice, to ensure adequate viral suppression, during the study.
    * Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
13. History of venous thrombosis within the past 3 months prior to the scheduled first dose of study treatment
14. Presence of acute coronary syndrome including myocardial infarction or unstable angina pectoris, other arterial thrombotic event including cerebrovascular accident or transient ischemic attack or stroke within the past 6 months prior to the scheduled first dose of study treatment
15. New York Heart Association (NYHA) Class II or greater congestive heart failure, serious cardiac arrhythmia requiring medication, or uncontrolled hypertension(more than 160 mmHg systolic and/or more than 100 mmHg diastolic, despite appropriate antihypertensive medication
16. Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab. The following are exceptions to this criterion:

    * Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
    * Systemic corticosteroids at physiologic doses not to exceed <<10 mg/day>> of prednisone or its equivalent
    * Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
17. Receipt of live attenuated vaccine within 30 days prior to the first dose of IP. Note: Patients, if enrolled, should not receive live vaccine whilst receiving IP and up to 30 days after the last dose of IP.
18. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab monotherapy.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-02-24 (Actual); Primary Completion 2023-03-09 (Actual); Study Completion 2023-03-09 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | 4 weeks
  To determine maximum tolerated dose of CKD-516 in combination with durvalumab

SECONDARY OUTCOMES:
To assess the safety and tolerability profile of CKD-516 in combination with Durvalumab | 1 year
  Adverse event according to NCI CTCAE v5.0
To assess the efficacy of CKD-516 in combination with Durvalumab; Objective Response | 1 year
  Objective Response Rate determined by Response Evaluation Criteria in Solid Tumors
Progression-free survival | 8 weeks
  - Progression free survival will be measured from the start of treatment with investigational product until the first documentation of disease progression or death due to any cause, whichever occurs first.
Duration of response | 1 year
  the duration from the first documentation of objective response to the first documented disease progression or death due to any cause, whichever occurs first
Overall survival | 1 year
  the time from the start of treatment with investigational product until death due to any cause.

OTHER OUTCOMES:
Translational biomarker assessments of tumor biopsy samples | 1 year
  TIL detected by multiplex IHC, Immunohistochemistry of SMAD4, STAT3
Translational biomarker assessments obtained from blood | 1 year
  Immune related-cytokine panel assay, Immune cell phenotyping

CONTACTS AND LOCATIONS:
Overall Officials: Tea Won Kim, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, Songpa-gu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alexandrov LB, Nik-Zainal S, Wedge DC, Aparicio SA, Behjati S, Biankin AV, Bignell GR, Bolli N, Borg A, Borresen-Dale AL, Boyault S, Burkhardt B, Butler AP, Caldas C, Davies HR, Desmedt C, Eils R, Eyfjord JE, Foekens JA, Greaves M, Hosoda F, Hutter B, Ilicic T, Imbeaud S, Imielinski M, Jager N, Jones DT, Jones D, Knappskog S, Kool M, Lakhani SR, Lopez-Otin C, Martin S, Munshi NC, Nakamura H, Northcott PA, Pajic M, Papaemmanuil E, Paradiso A, Pearson JV, Puente XS, Raine K, Ramakrishna M, Richardson AL, Richter J, Rosenstiel P, Schlesner M, Schumacher TN, Span PN, Teague JW, Totoki Y, Tutt AN, Valdes-Mas R, van Buuren MM, van 't Veer L, Vincent-Salomon A, Waddell N, Yates LR; Australian Pancreatic Cancer Genome Initiative; ICGC Breast Cancer Consortium; ICGC MMML-Seq Consortium; ICGC PedBrain; Zucman-Rossi J, Futreal PA, McDermott U, Lichter P, Meyerson M, Grimmond SM, Siebert R, Campo E, Shibata T, Pfister SM, Campbell PJ, Stratton MR. Signatures of mutational processes in human cancer. Nature. 2013 Aug 22;500(7463):415-21. doi: 10.1038/nature12477. Epub 2013 Aug 14. PMID 23945592
- [Background] Brahmer JR, Tykodi SS, Chow LQ, Hwu WJ, Topalian SL, Hwu P, Drake CG, Camacho LH, Kauh J, Odunsi K, Pitot HC, Hamid O, Bhatia S, Martins R, Eaton K, Chen S, Salay TM, Alaparthy S, Grosso JF, Korman AJ, Parker SM, Agrawal S, Goldberg SM, Pardoll DM, Gupta A, Wigginton JM. Safety and activity of anti-PD-L1 antibody in patients with advanced cancer. N Engl J Med. 2012 Jun 28;366(26):2455-65. doi: 10.1056/NEJMoa1200694. Epub 2012 Jun 2. PMID 22658128
- [Background] Brem S, Brem H, Folkman J, Finkelstein D, Patz A. Prolonged tumor dormancy by prevention of neovascularization in the vitreous. Cancer Res. 1976 Aug;36(8):2807-12. PMID 1277191
- [Background] Butte MJ, Keir ME, Phamduy TB, Sharpe AH, Freeman GJ. Programmed death-1 ligand 1 interacts specifically with the B7-1 costimulatory molecule to inhibit T cell responses. Immunity. 2007 Jul;27(1):111-22. doi: 10.1016/j.immuni.2007.05.016. Epub 2007 Jul 12. PMID 17629517
- [Background] Comunanza V, Bussolino F. Therapy for Cancer: Strategy of Combining Anti-Angiogenic and Target Therapies. Front Cell Dev Biol. 2017 Dec 7;5:101. doi: 10.3389/fcell.2017.00101. eCollection 2017. PMID 29270405
- [Background] Dong C, Li Z, Alvarez R Jr, Feng XH, Goldschmidt-Clermont PJ. Microtubule binding to Smads may regulate TGF beta activity. Mol Cell. 2000 Jan;5(1):27-34. doi: 10.1016/s1097-2765(00)80400-1. PMID 10678166
- [Background] Dunn GP, Old LJ, Schreiber RD. The three Es of cancer immunoediting. Annu Rev Immunol. 2004;22:329-60. doi: 10.1146/annurev.immunol.22.012703.104803. PMID 15032581
- [Background] Ellis S, Carroll KJ, Pemberton K. Analysis of duration of response in oncology trials. Contemp Clin Trials. 2008 Jul;29(4):456-65. doi: 10.1016/j.cct.2007.10.008. Epub 2007 Nov 12. PMID 18187370
- [Background] Fife BT, Bluestone JA. Control of peripheral T-cell tolerance and autoimmunity via the CTLA-4 and PD-1 pathways. Immunol Rev. 2008 Aug;224:166-82. doi: 10.1111/j.1600-065X.2008.00662.x. PMID 18759926
- [Background] Hirano F, Kaneko K, Tamura H, Dong H, Wang S, Ichikawa M, Rietz C, Flies DB, Lau JS, Zhu G, Tamada K, Chen L. Blockade of B7-H1 and PD-1 by monoclonal antibodies potentiates cancer therapeutic immunity. Cancer Res. 2005 Feb 1;65(3):1089-96. PMID 15705911
- [Background] Hori K, Saito S. Microvascular mechanisms by which the combretastatin A-4 derivative AC7700 (AVE8062) induces tumour blood flow stasis. Br J Cancer. 2003 Oct 6;89(7):1334-44. doi: 10.1038/sj.bjc.6601261. PMID 14520469
- [Background] Iwai Y, Ishida M, Tanaka Y, Okazaki T, Honjo T, Minato N. Involvement of PD-L1 on tumor cells in the escape from host immune system and tumor immunotherapy by PD-L1 blockade. Proc Natl Acad Sci U S A. 2002 Sep 17;99(19):12293-7. doi: 10.1073/pnas.192461099. Epub 2002 Sep 6. PMID 12218188
- [Background] Keir ME, Butte MJ, Freeman GJ, Sharpe AH. PD-1 and its ligands in tolerance and immunity. Annu Rev Immunol. 2008;26:677-704. doi: 10.1146/annurev.immunol.26.021607.090331. PMID 18173375
- [Background] Lu Y, Chen J, Xiao M, Li W, Miller DD. An overview of tubulin inhibitors that interact with the colchicine binding site. Pharm Res. 2012 Nov;29(11):2943-71. doi: 10.1007/s11095-012-0828-z. Epub 2012 Jul 20. PMID 22814904
- [Background] Fens MH, Storm G, Schiffelers RM. Tumor vasculature as target for therapeutic intervention. Expert Opin Investig Drugs. 2010 Nov;19(11):1321-38. doi: 10.1517/13543784.2010.524204. Epub 2010 Oct 15. PMID 20946091
- [Background] Kamran MZ, Patil P, Gude RP. Role of STAT3 in cancer metastasis and translational advances. Biomed Res Int. 2013;2013:421821. doi: 10.1155/2013/421821. Epub 2013 Oct 2. PMID 24199193
- [Background] Narwal R, Roskos LK, Robbie GJ. Population pharmacokinetics of sifalimumab, an investigational anti-interferon-alpha monoclonal antibody, in systemic lupus erythematosus. Clin Pharmacokinet. 2013 Nov;52(11):1017-27. doi: 10.1007/s40262-013-0085-2. PMID 23754736
- [Background] Ng CM, Lum BL, Gimenez V, Kelsey S, Allison D. Rationale for fixed dosing of pertuzumab in cancer patients based on population pharmacokinetic analysis. Pharm Res. 2006 Jun;23(6):1275-84. doi: 10.1007/s11095-006-0205-x. Epub 2006 May 26. PMID 16715358
- [Background] Okudaira K, Hokari R, Tsuzuki Y, Okada Y, Komoto S, Watanabe C, Kurihara C, Kawaguchi A, Nagao S, Azuma M, Yagita H, Miura S. Blockade of B7-H1 or B7-DC induces an anti-tumor effect in a mouse pancreatic cancer model. Int J Oncol. 2009 Oct;35(4):741-9. doi: 10.3892/ijo_00000387. PMID 19724910
- [Background] Pardoll DM. The blockade of immune checkpoints in cancer immunotherapy. Nat Rev Cancer. 2012 Mar 22;12(4):252-64. doi: 10.1038/nrc3239. PMID 22437870
- [Background] Paterson AM, Brown KE, Keir ME, Vanguri VK, Riella LV, Chandraker A, Sayegh MH, Blazar BR, Freeman GJ, Sharpe AH. The programmed death-1 ligand 1:B7-1 pathway restrains diabetogenic effector T cells in vivo. J Immunol. 2011 Aug 1;187(3):1097-105. doi: 10.4049/jimmunol.1003496. Epub 2011 Jun 22. PMID 21697456
- [Background] Pilat MJ, Lorusso PM. Vascular disrupting agents. J Cell Biochem. 2006 Nov 1;99(4):1021-39. doi: 10.1002/jcb.20783. PMID 16927308